CLINICAL TRIAL: NCT00508274
Title: An Open-Label Multicenter Study Administering Lapatinib and Capecitabine (Xeloda) in Women With Advanced or Metastatic Breast Cancer
Brief Title: Lapatinib +Capecitabine Treatment for Advanced Metastatic Breast Cancer in Women From China
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary analysis was completed in 2015 and data collection post 1-Jul-2019 was not reportable due to local regulations in China.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF109491; CLAP016A2304 (Other: Novartis)
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Results first posted 2009-09-03 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Neoplasms, Breast
Keywords: Advanced Metastatic Breast Cancer; HER2 positive; HER2+; breast cancer; lapatinib; TYVERB; TYKERB; Capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lapatinib in combination with capecitabine (Experimental): daily oral lapatinib (1250 mg/day) in combination with capecitabine (2000mg/m2/day on days1-14 every 21 days)
  Interventions: Drug: lapatinib; Drug: capecitabine

INTERVENTIONS:
Drug: lapatinib — Lapatinib ditosylate monohydrate tablets, 250 mg, are oval, biconvex, orange, film-coated tablets taken orally.
  Other Names: LAP016, GW572016
Drug: capecitabine — Capecitabine is supplied as a biconvex, oblong, light peach and peach colored, film-coated tablets for oral administration.

SUMMARY:
Local study in China and Hong Kong to evaluate safety and efficacy in lapatinib + capecitabine in women with Human epidermal growth factor receptor 2 (HER2) positive advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
The Primary objective of the study was to evaluate the overall clinical benefit response (CBR) rate.

This was a single arm, open-label, multi-center study of lapatinib plus capecitabine in women from mainland China and Hong Kong who had advanced or metastatic breast cancer that progressed on prior chemotherapies with or without trastuzumab.

Participants received study treatment until disease progression, unacceptable toxicity, or withdrawal for any other reasons.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Female ≥18 years;
* Pathology that has histologically confirmed invasive breast cancer with stage IIIb/c or stage IV disease;

  • If recurrent disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology or histology.
* Documented overexpression of Her2 (ErbB2) of IHC 3+ or FISH positive, in primary or metastatic tumor tissue is required for enrollment into the study; by local testing or central laboratory testing determined by country of residence. NB. Approximately, 51 subjects will be enrolled in a single stage design to test for efficacy in women from China and Hong Kong. Due to the fact that trastuzumab is not commonly prescribed in China and Hong Kong, the current study allows up to 40% of subjects who are trastuzumab naïve to be enrolled.
* Prior therapies must include at minimum a taxane and/or anthracycline and may include trastuzumab if available; other prior regimens are not limited except capecitabine and Erbb2 inhibitors other than trastuzumab. Chemo regimen requirements are as follows:

  * Taxane containing regimen for at least 4 cycles or <4 cycles provided disease progression or treatment limiting toxicity occurred while on taxane
  * Anthracycline containing regimen for at least 4 cycles or <4 cycles provided disease progression or treatment limiting toxicity occurred while on anthracycline
  * Taxanes and Anthracyclines may have been administered concurrently or separately
  * Prior treatment may have contained trastuzumab alone or in combination with other chemotherapy in the adjuvant, locally advanced or metastatic setting and patient must have failed the treatment
  * Prior treatment with capecitabine is not permitted unless 6 months have elapsed since the last dose of capecitabine and the subject is free of any capecitabine related toxicity
  * Prior therapy with an ErbB1 and/or ErbB2 inhibitor, other than trastuzumab is not permitted
  * Other prior chemo-regimens not listed above are unlimited.
* For those subjects whose disease is ER+ and/or PR+ one of following criteria should be met.

  * Subjects who received hormonal therapy and are no longer benefiting from this therapy and the hormonal treatment must have been stopped before the first dose of investigational treatment
  * Subjects with visceral disease that requires chemotherapy (eg., subjects with liver or lung metastases)
  * Rapidly progressing or life threatening disease, as determined by the investigator
* Subjects with stable CNS metastases (asymptomatic and off systemic steroids and anticonvulsants for at least 3 months) are eligible
* Measurable lesion(s) according to RECIST (Response Evaluation Criteria in Solid Tumors);
* Radiotherapy as palliative treatment for painful metastatic disease is permitted but must have been stopped within 2 weeks prior to initiation of any investigational treatment. All subjects must have recovered from all radiotherapy related toxicities prior to initiation of any investigational treatment. The site of radiotherapy must not be used as a site of measurable disease;
* Cardiac ejection fraction within institutional range of normal as measured by echocardiogram. MUGA scans will be accepted in cases where an echocardiogram cannot be performed or is inconclusive;
* ECOG Performance Status of 0 to 1;
* Life expectancy of ≥ 12 weeks;
* Able to swallow and retain oral medication;
* Women with potential to have children must be willing to practice acceptable methods of birth control during the study;
* Willing to complete all screening assessments as outlined in the protocol;
* Adequate organ function as defined by the Table of Baseline Laboratory Values

Exclusion Criteria:

* Pregnant or lactating females at anytime during the study
* Subjects with only non-measurable metastatic sites of disease per RECIST, (e.g. bone metastases, pleural effusion, or ascites, etc.);
* Planned concurrent anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy) while taking investigational treatment;
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded;
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible;
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety;
* Uncontrolled infection;
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-07-18 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- China (6):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Shatin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Xu BH, Jiang ZF, Chua D, Shao ZM, Luo RC, Wang XJ, Liu DG, Yeo W, Yu SY, Newstat B, Preston A, Martin AM, Chi HD, Wang L. Lapatinib plus capecitabine in treating HER2-positive advanced breast cancer: efficacy, safety, and biomarker results from Chinese patients. Chin J Cancer. 2011 May;30(5):327-35. doi: 10.5732/cjc.010.10507. PMID 21527065

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib + Capecitabine: Daily oral lapatinib (1250 mg/day) in combination with capecitabine (2000 mg/m2/day on Days 1-14 every 21 Days); m2 = Square meter: Body Surface Area
Period: Overall Study
Arm/Group | Lapatinib + Capecitabine
Started | 52
Completed | 2
Not Completed | 50
Not completed — Adverse Event | 5
Not completed — Death | 7
Not completed — Disease progression | 32
Not completed — Withdrawal by Subject | 1
Not completed — Subject received new anti-cancer chemotherapy/traditional Chinese medicine | 2
Not completed — Missing | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 52

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined by the percentage of participants achieving either a confirmed tumor response of complete response (CR) or partial response (PR) or stable disease (SD) for at least 24 weeks. Response Criteria in Solid Tumors (RECIST) is a system for measuring tumor shrinkage or progression in terms of the longest dimensions of the tumor on imaging scans such as computerized tomography (CT). A "partial response" requires a decrease of 30% or more, "complete response" requires all target lesions disappear, "Progression" requires an increase of at least 20%, and "Stable disease" falls in between these two. All responses have a repeat assessment to confirm the response.
Time Frame: Baseline; every 6 weeks for the first 36 weeks and then every 12 weeks until disease progression. The maximum time participants were followed was approx. 90 months
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of investigational product
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 52
Percentage of participants | 57.7 [43.2 to 71.3]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from first dose date until the date of disease progression or death due to any reason, whichever occurs first.
Time Frame: Baseline; every 6 weeks for the first 36 weeks and then every 12 weeks until disease progression. The maximum time participants were followed was 90.38 months.
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of investigational product
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 52
Months | 6.34 [0.03 to 90.38]

3. Secondary Outcome: Six Months Progression-Free Survival
Description: Six Months Progression-Free Survival is defined as the percentage of surviving participants who are progression-free longer than six months (greather than 180 days) after the first start date of study treatment.
Time Frame: at Baseline and every 6 weeks for the first 36 weeks and then every 12 weeks until disease progression. The maximum time participants were followed up to 90.38 months, with 6 months PFS reported.
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of investigational product
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 52
Percentage of participants | 53.55 [38.77 to 66.25]

4. Secondary Outcome: Time to Response (TTR)
Description: Time to response is defined as the time from first dose date until first documentation of disease response. TTR only applied to participants for whom best overall response was complete response (CR), partial response (PR) or stable disease (SD). Participants who had not had a partial response, complete response or stable disease at the cut-off date for this endpoint analysis were censored for time to response.
Time Frame: Baseline; every 6 weeks for the first 36 weeks and then every 12 weeks until disease progression. The maximum time participants were followed was approx. 14.78 months
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of investigational product. TTR only applied to participants for whom best overall response was complete response (CR) or partial response (PR) or stable disease.
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 23
Months | 4.07 [2.73 to 14.78]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (complete response, partial response or stable disease) is defined as the time of first documentation of disease response until the date of disease progression or death due to breast cancer, whichever occurs first. DOR only applied to participants for whom best overall response was complete response (CR), partial response (PR) or stable disease (SD). Participants who had not had a partial response, complete response or stable disease at the cut-off date for this endpoint analysis were censored for duration of response.
Time Frame: Baseline; every 6 weeks for the first 36 weeks and then every 12 weeks until disease progression. The maximum time participants were followed was 88.80 months.
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of investigational product. DOR only applied to participants for whom best overall response is complete response (CR) or partial response (PR) or stable disease (SD).
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 23
Months | 8.18 [2.69 to 88.80]

6. Secondary Outcome: Number of Participants With Central Nervous System (CNS) as First Site of Relapse
Description: Number of participants who had Central Nervous System metastasis as the first site of relapse. CT, Magnetic Resonance Imaging, etc. were used for the assessment.
Time Frame: Baseline; every 6 weeks for the first 36 weeks and then every 12 weeks until disease progression. The maximum time participants were followed was 90 months
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of investigational product
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 52
participants
  Participants with any site of relapse | 17
  Participants with CNS disease as first site of relapse | 2

7. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from the start of treatment up to 30 days after study drug discontinuation, for a maximum duration of 4276 days (treatment duration ranged from 13 - 4246 days) for Lapatinib and 3384 days (treatment duration ranged form 8 - 3354 days) for Capecitabine. Total deaths was collected from study start to study end (LPLV).
Time Frame: up to 4276 days for Lapatinib/up to 3384 days for Capecitabine (on-treatment), approx. 12 years (all collected deaths)
Population: Clinical Database Population: all treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 52
Participants
  Total Deaths | 11
  On-treatment Deaths | 2

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 4276 days for Lapatinib, including the 30 days safety follow- up (treatment duration ranged from 13 to 4246 days) and 3384 days for Capecitabine, including the 30 days safety follow up (treatment duration ranged from 8 to 3354 days).
Description: AE: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Arm/Group | Lapatinib + Capecitabine
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 4/52
Other Adverse Events (participants affected / at risk) | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Capecitabine (N=52)
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaginal Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Capecitabine (N=52)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 26
Mouth Ulceration (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 3
Fatigue (General disorders) | 13
Pyrexia (General disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 20
Liver Injury (Hepatobiliary disorders) | 4
Alanine Aminotransferase Increased (Investigations) | 4
Aspartate Aminotransferase Increased (Investigations) | 4
Blood Bilirubin Increased (Investigations) | 5
Neutrophil Count Decreased (Investigations) | 3
White Blood Cell Count Decreased (Investigations) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 32
Rash (Skin and subcutaneous tissue disorders) | 26

LIMITATIONS AND CAVEATS:
Data collection post 1-Jul-2019 was not reportable due to local regulations in China.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety